CLINICAL TRIAL: NCT02493543
Title: Role of Autoantibodies in Spontaneous Functional Recovery After Spinal Cord Injury
Brief Title: Autoantibodies on Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital Nacional de Parapléjicos de Toledo (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Principal Investigator, Dr. Angel Arevalo Martin, Ph.D., Hospital Nacional de Parapléjicos de Toledo
Other Study IDs: FMM14
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Spinal Cord Injuries
Keywords: autoantibodies
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Spinal cord injury: Patients (n=90) will undergo a common arm blood collection to determine autoantibody profiles in serum. This procedure will be performed twice: after recruitment and 3 months later.
  Interventions: Other: Blood collection
- Controls: Control subjects (n=20) will undergo a common arm blood collection to determine autoantibody profiles in serum. This procedure will be performed only once.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Blood collection from the subject's arm

SUMMARY:
The purpose of this study is to determine the autoantibody profiles after spinal cord injury and their role in spontaneous functional recovery.

DETAILED DESCRIPTION:
Most patients experience variable degrees of functional recovery after spinal cord injury (SCI), predominantly in the first months after lesion. In SCI animal models, autoantibodies are pathogenic and their titers rise up at the time when spontaneous recovery stops. The aim of this study is to determine the autoantibody profiles after SCI and to infer their relation with functional recovery. To achieve this, autoantibody profiles, biochemical, hematological and immune-related parameters (cytokines, chemokines and growth factors) will be determined from a serum blood sample and functional recovery will be evaluated accordingly to standardized scales.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic or non-progressive vascular SCI
* Less than 45 days after lesion
* Any neurological level
* Complete and incomplete lesions
* If patient has been treated with glucocorticoids, it should have passed at least 7 days from the end of the treatment

Exclusion Criteria:

* Cauda equina syndrome
* Autoimmune disorder
* Tumor (even if benign)
* Neurodegenerative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute spinal cord injury admitted to the Spanish National Hospital for Paraplegics
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2014-10-17 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Changes in ASIA scores | 4 months

SECONDARY OUTCOMES:
Change in neurological level of injury | 4 months
Change in ASIA impairment scale (AIS) | 4 months

OTHER OUTCOMES:
Spinal cord independence measure (SCIM) | Until discharge from the hospital (6-12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Angel Arevalo-Martin, PhD, Principal Investigator — Hospital Nacional de Parapléjicos, SESCAM
Locations (2):
- Berufsgenossenschaftliche Unfallklinik Murnau, Murnau am Staffelsee, Germany
- Hospital Nacional de Parapléjicos, SESCAM, Toledo, Spain

REFERENCES:
- [Derived] Leister I, Altendorfer B, Maier D, Mach O, Wutte C, Grillhosl A, Arevalo-Martin A, Garcia-Ovejero D, Aigner L, Grassner L. Trajectory of Serum Levels of Glial Fibrillary Acidic Protein Within Four Weeks Post-Injury Is Related to Neurological Recovery During the Transition from Acute to Chronic Spinal Cord Injury. J Neurotrauma. 2023 May;40(9-10):999-1006. doi: 10.1089/neu.2022.0326. Epub 2022 Dec 9. PMID 36200629